CLINICAL TRIAL: NCT03466840
Title: Clinical Assessment of Coronally Advanced Lingual Flap to Modified Periosteal Releasing Incision for Flap Advancement in Partially Edentulous Patients Undergoing Guided Bone Regeneration Using Titanium Mesh.
Brief Title: Comparison of Coronally Advanced Lingual Flap to Modified MPI for Flap Advancement in Partially Edentulous Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Fathi Messalam Diab, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cebc. cairouniversity
Record Dates: First submitted 2018-01-11; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Alveolar Bone Loss
Keywords: Ridge Augmentation; Titanium mesh; Flap advancement
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant
Masking Description: According to the allocation sequence obtained from the computer software the numbers will be written in small folded opaque papers and put in opaque sealed envelopes. All those papers will be ready before conducting any procedure. The patients will be allowed to pick his/her number from the pile of envelopes and will be assigned accordingly. The number of papers will decrease as each patient picks his number and so on.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Coronally Advanced Lingual Flap (Experimental): On the lingual side of mandible, a full-thickness muco-periosteal flap is elevated until reaching mylohyoid line. Using a blunt instrument, a connective tissue band is localized continuing with the epimysium of the mylohyoid muscle and is inserted into the inner part of the lingual flap . The blunt instrument is inserted below the connective band, and with gentle traction in the coronal direction, this muscular insertion was detached from the lingual flap. Using a "periodontal probe" the amount of advancement is measured.
  Interventions: Procedure: The coronally advanced lingual flap
- Modified periosteal releasing Incision (Active Comparator): A full-thickness muco-periosteal flap is reflected on the buccal side. Near the base of muco-periosteal flap, the periosteum is incised less than 0.5mm in depth, creating two segments, "coronal segment" and "apical segment," of the periosteal flap. The flap is pulled with a pair of periodontal forceps laterally. Subsequently, the "lateral stretching" of the coronal segment of the flap is performed by applying pressure using the blunt face of scalpel blade, or a blunt instrument, with sweeping motion. This motion helps stretching the flap over the submucosa, thereby permitting the flap to be mobile.Using a "periodontal probe" the amount of advancement is measured
  Interventions: Procedure: Modified periosteal releasing Incision

INTERVENTIONS:
Procedure: The coronally advanced lingual flap — : A full-thickness crestal incision is performed from the distal surface of the more distal tooth to retromolar pad and finishing with releasing incision. On the lingual side, a full-thickness muco-periosteal flap was elevated until reaching mylohyoid line. Then using a blunt instrument, it was localized a connective tissue band continuing with the epimysium of the mylohyoid muscle. It is inserted into the inner part of the lingual flap about 5mm from the crest in an apical direction. The blunt instrument is inserted below the connective band, and with gentle traction in the coronal direction, this muscular insertion was detached from the lingual flap. Using a "periodontal probe", the amount of advancement is measured.
  Arms: The Coronally Advanced Lingual Flap
Procedure: Modified periosteal releasing Incision — A full-thickness muco-periosteal flap is reflected on the buccal side. Near the base of muco-periosteal flap, the periosteum is incised less than 0.5mm in depth, creating two segments, "coronal segment" and "apical segment," of the periosteal flap. The flap is pulled with a pair of periodontal forceps laterally. Subsequently, the "lateral stretching" of the coronal segment of the flap is performed by applying pressure using the blunt face of scalpel blade, or a blunt instrument, with sweeping motion. This motion helps stretching the flap over the submucosa, thereby permitting the flap to be mobile.Using a "periodontal probe" the amount of advancement is measured.
  Arms: Modified periosteal releasing Incision

SUMMARY:
Comparison of cronally advanced lingual flap to modified periosteal releasing incision (MPRI)

DETAILED DESCRIPTION:
Clinical Assessment and Comparison of Coronally Advanced Lingual Flap to Modified Periosteal Releasing Incision for Flap Advancement in Partially Edentulous Patients Undergoing Guided Bone Regeneration Using Titanium Mesh: A Randomized Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous patients in the mandibular posterior region.
* Patients with healthy systemic condition.
* Insufficient ridge width (< 5mm).
* Presence of proper inter-arch space for placement of the implant prosthetic part.
* Adequate soft tissue biotype (≥ 2 mm).

Exclusion Criteria:

* Patients with systemic conditions that may interfere with the results of the study.
* Patients with local pathological defects related to the area of interest.
* Unmotivated, uncooperative patients with poor oral hygiene.
* Patients with habits that may jeopardize the implant longevity and affect the results of the study such as smoking, alcoholism or para-functional habits.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-08-25 (Estimated)

PRIMARY OUTCOMES:
Flap advancement | "10 minutes"
  Flap advancement will be measured as a difference between the value before and after in millimeters using periodontal probe.

SECONDARY OUTCOMES:
Postoperative Pain | 1 Week
  Postoperative Pain will be recorded using Numerical Rating scale (NRS) The scores will be recorded postoperatively by the patient for the seven days of observation.
Postoperative membrane exposure | 12 Weeks
  Postoperative membrane exposure will be evaluated at 1, 2, 3, 4, 12 weeks using a periodontal probe in millimeters.
bone density | 12 Weeks
  bone density will before and after with cone beam computed tomography (CBCT)
postoperative swelling | "1 week"
  postoperative swelling will be recorded using descriptive four point scale(Penarrocha et al.2006).The scores will be recorded postoperatively by the patient for the seven days of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Egypt Recruiting, Principal Investigator — Cairo, Egypt, 02
Locations (1):
- Noha Diab, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided